CLINICAL TRIAL: NCT06694779
Title: Thrombosis in Diffuse Large B-cell Lymphoma: Impact on Outcome, Evaluation, and Comparison of Predictive Models of Thrombotic Risk: Multicentre Retrospective Observational Study. the PREDIC-TO (PREDICt ThrOmbosis) Study
Brief Title: Thrombosis in Diffuse Large B-cell Lymphoma:the PREDIC-TO (PREDICt ThrOmbosis) Study
Acronym: PREDIC-TO
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: PREDIC-TO
Record Dates: First submitted 2023-07-17; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Large B Cell Lymphoma; Thrombosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Comparative Evaluation of Thrombotic Risk Models in DLBCL patients

Objective: To assess the impact of thrombotic risk factors and compare the performance of existing predictive models (Khorana, Throly, Model IX) in Diffuse Large B-cell Lymphoma (DLBCL)

Primary Endpoints:

Measure thrombotic risk factors in existing models Determine occurrence, type, and timing of venous thrombotic events

Secondary Endpoints:

Assess performance of models in patients without thrombotic events at diagnosis Evaluate dynamic risk factors during DLBCL treatment Identify additional risk factors not included in published models Analyze overall survival and VTE-free survival

Methodology:

Real-world cohort study of DLBCL patients Collection of static and dynamic risk factors Correlation analysis of risk factors with thrombotic events Development and validation of DLBCL-specific predictive model

Conclusion:

This study aims to compare existing predictive models and develop a DLBCL-specific model to aid in identifying high-risk patients and inform thromboprophylaxis decisions. Results will contribute to improved understanding and management of thrombotic risk in DLBCL.

DETAILED DESCRIPTION:
DLBCL is the most frequent lymphoid malignancy in the adult population and the one with the highest risk of thrombotic events. The indications for thromboprophylaxis are, however, debated.

For such reason, risk scores (i.e., the Khorana, Throly and the recently published Model IX score), have been developed to identify patients bearing a high thrombotic risk at diagnosis. These models, however, were developed considering not only aggressive lymphomas, but also indolent lymphomas, characterized by a markedly lower risk of VTE when compared to DLBCL.

The performance of the Khorana, Throly and Model IX score has never been evaluated and compared in the sole DLBCL population. Such understanding in a cohort of "real world" patients could aid clinicians in deciding whether to initiate thromboprophylaxis and may direct randomised controlled trials on the use of prophylactic heparin in the future.

Moreover, the aforementioned scores assess independent variables at diagnosis, not taking into account the possible occurrence of risk factors that may arise over the course of DLBCL treatment or in case of placement of a central venous catheter (CVC).

Assessing the impact of thrombotic risk factors at diagnosis and during the disease, in a cohort of sole DLBCL patients, could allow the development of a new predictive model of thrombotic risk adapted to DLBCL.

5. OBJECTIVES AND ENDPOINTS OBJECTIVES Primary objective

- To assess the impact of thrombotic risk factors on the development of VTE in patients with Diffuse Large B-cell Lymphoma (DLBCL): real-life comparison of models predictive of thrombotic risk (Khorana, Throly and Model IX scores).

Secondary objectives

* To evaluate the statistical performance of the aforementioned predictive models in the subgroup of patients who did not have a thrombotic event at diagnosis
* To assess the impact of dynamic risk factors (i.e., not present at diagnosis) on thrombotic risk
* To evaluate the impact of risk factors at diagnosis which are not included in the published predictive models
* To evaluate overall survival and VTE-free survival
* Creation of a predictive model of thrombotic risk adapted to DLBCL

ENDPOINTS Primary endpoints

* Measurement of thrombotic risk factors present in the Khorana, Throly and Model IX scores: previous arterial or venous thrombotic event, ECOG, weight, extra nodal and/or mediastinal localization of disease, leukocytes, neutrophils, haemoglobin, platelet count, albumin, bulky mass
* Occurrence of arterial and venous thrombotic events, type of event, time to event after diagnosis and during disease

Secondary endpoints

* Data collection of static thrombotic risk factors at diagnosis and not included in the already published scores:

  * de novo or secondary DLBCL status
  * Neutrophil/lymphocyte ratio (ANC/ALC ratio)
  * Cardio aspirin
  * R-IPI
  * Immunohistochemistry: Ki67, Myc, CD10, BCL-6, BCL-2
* Correlation between static risk factors at diagnosis and relative risk of thrombotic events
* Data collection of dynamic risk factors (as both categorical-dichotomous and temporal variable) present from diagnosis to expected event, death or lost at follow-up:

  * Central venous catheter placement
  * Therapy: radiotherapy, chemotherapy, anthracycline therapy, number of therapeutic lines, autologous haematopoietic stem cell transplantation
  * LDH, haemoglobin < 10 g/dl if > than 10 at diagnosis, venous compression at CT scan, extra nodal localisation if not present at diagnosis, albumin < 3.5 g/dl if greater at diagnosis
  * ANC/ALC ratio at the time of thrombotic event
* Correlation between acquisition of dynamic risk factors and relative risk of thrombotic event
* Date of thrombotic event, death or lost to follow-up to determine overall survival and VTE free survival
* Creation and validation of a predictive model adapted to DLBCL based on the Hazard Ratios of the independent variables

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥ 18 years
* Histological diagnosis of DLBCL
* Informed consent freely given and obtained

Exclusion Criteria:

* Active anticoagulant therapy at the time of diagnosis
* Start of prophylactic heparin following diagnosis
* Absence of necessary data to extrapolate risk scores (Khorana, Throly and Model IX) at diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -. Patients with a diagnosed of DLBCL from 01/01/2004 until 31/12/2022 can be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Measurement of thrombotic events | From the date of diagnosis of Diffuse Large B-Cell Lymphoma (DLBCL) to the occurrence of a thrombotic event (arterial or venous), death, loss to follow-up, or a maximum period of 24 months from diagnosis, whichever comes first.
  Measurement of thrombotic risk factors present in the Khorana, Throly and Model IX scores.
  Thrombotic events after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ivan Civettini, Monza, Italy, Italy

IPD SHARING:
Plan to Share IPD: No